CLINICAL TRIAL: NCT06641401
Title: A Case Series of Endoscopic Flexor Hallucis Longus Transfer for Acute Achilles Tendon Rupture.
Brief Title: Endoscopic FHL Transfer for Acute Achilles Tendon Rupture
Status: Enrolling by invitation | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: General Hospital of Naoussa (Unknown)
Responsible Party: Principal Investigator, Michail Kotsapas, Michail Kotsapas, MD, MSc, Resident of Orthopedics (General Hospital of Naoussa), PhD Candidate (Aristotle University of Thessaloniki), Aristotle University Of Thessaloniki
Other Study IDs: 6/14.6.2022
Record Dates: First submitted 2024-10-12; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Achilles Tendon Rupture; Achilles Tendon Injury; Achilles Tendon Surgery; Flexor Hallucis Longus
Keywords: Achilles tendon, rupture, endoscopic, flexor hallucis longus transfer
MeSH Terms: conditions — Rupture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endoscopic Flexor Hallucis Longus Transfer Group: 28 Patients with acute Achilles tendon rupture treated with Endoscopic Flexor Hallucis Longus transfer by a single surgeon in a single hospital (General Hospital of Naousa, Greece). All patients followed the same postoperative rehabilitation program.
  Interventions: Procedure: Endoscopic Flexor Hallucis Longus transfer for Acute Achilles tendon rupture

INTERVENTIONS:
Procedure: Endoscopic Flexor Hallucis Longus transfer for Acute Achilles tendon rupture — All patients have already undergone the same operation for the same disease. All data are to be collected retrospectively

SUMMARY:
This observational study aims to evaluate the outcome of endoscopic flexor hallucis longus transfer (FHLt) in patients with acute Achilles tendon rupture (AATR).

DETAILED DESCRIPTION:
This evaluation will be performed by examining the following parameters:

1. Patient satisfaction quantified with the Achilles tendon Total Rupture Score (ATRS). This is the primary outcome.
2. Complication rate
3. Ankle and Calf circumference compared to the contralateral healthy limb.
4. Passive and Active range of ankle motion compared to the contralateral healthy limb.
5. Hallux flexion force compared to the contralateral healthy limb.

ELIGIBILITY:
Inclusion Criteria:

* Signed Consent Form
* Acute Achilles Tendon Rupture (<4 weeks)
* Underwent operative treatment with Endoscopic Flexor Hallucis Longus transfer
* More than 24 months postoperative follow-up
* Patients operated after 2015

Exclusion Criteria:

* Inability or Unwillingness to cooperate
* Medically unfit for examination
* Age less than 18 or more than 75 years
* Non-operative Management or any other Surgical Management
* Neglected Achilles Tendon Rupture (>4 weeks)
* Bilateral Achilles Tendon Rupture
* Patients operated before 1.1.2015 or after 1.1.2023
* Comorbidities interfering with the secondary outcomes (e.g. Venous insufficiency resulting in lower limb excessive edema interferes with ankle and calf circumference, rheumatoid arthritis and/or previous foot and ankle surgery interferes with active and passive range of motion of the ankle, etc)

Ages: 18 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who underwent endoscopic flexor hallucis longus transfer for acute Achilles tendon rupture by a single surgeon in a single hospital
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2023-03-05 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction | At least 24 months postoperatively
  Evaluated and quantified with the Achilles Tendon Total Rupture Score (min = 0 - worst outcome, max = 100 - best outcome)

SECONDARY OUTCOMES:
Complication rate | At least 24 months postoperatively
  Complications will be recorded and categorized: Rerupture, Infection, Nerve injury, Miscellaneous
Calf Circumference | At least 24 months postoperatively
  Calf circumference measured 15 cm distally to the inferior pole of the patella. Contralateral limb calf circumference will also be measured. The Calf Circumference Difference will be calculated and compared between the two groups.
Ankle Circumference | At least 24 months postoperatively
  Ankle circumference measured 8 cm proximally to the lateral malleolus. Contralateral limb ankle circumference will also be measured. The Ankle Circumference Difference will be calculated and compared between the two groups.
Ankle Range of Motion | At least 24 months postoperatively
  Active and Passive Ankle joint Range of Motion will be calculated with an electronic goniometer. Contralateral limb Range of Ankle joint Motion will also be measured. The Range of Motion Difference will be calculated and compared between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Michail Kotsapas, MD, MSc, Principal Investigator — General Hospital of Naousa, Department of Orthopedics
Locations (1):
- General Hospital of Naousa, Náousa, Central Macedonia, Greece

IPD SHARING:
Plan to Share IPD: Undecided
The records of each patient to be enrolled belong to the General Hospital of Naousa. The records of each patient will be entrusted to the main researcher (M.K.) with the obligation to maintain doctor-patient confidentiality. The final study results will not reveal any sensitive patient data (de-identification). Photos and videos of each patient's examination may be taken after ensuring their written and oral informed consent.

REFERENCES:
- [Background] Abdelatif NMN, Batista JP. Endoscopic Flexor Hallucis Longus Transfer for the Management of Acute Achilles Tendon Ruptures in Professional Soccer Players. Foot Ankle Int. 2022 Feb;43(2):164-175. doi: 10.1177/10711007211036439. Epub 2021 Sep 24. PMID 34558318
- [Result] Batista JP, Abdelatif NMN, Del Vecchio JJ, Diniz P, Pereira H. Endoscopic Flexor Hallucis Longus Transfer for the Management of Acute Achilles Tendon Ruptures: A Prospective Case Series Report With a Minimum of 18 Months' Follow-Up. J Foot Ankle Surg. 2020 Sep-Oct;59(5):927-937. doi: 10.1053/j.jfas.2019.12.008. Epub 2020 Jun 9. PMID 32527698